CLINICAL TRIAL: NCT04826289
Title: Radiological Assessment of Vertical Distance Between Medial and Lateral Malleolus in Normal Population
Brief Title: Vertical Distance Between Medial and Lateral Malleolus in Normal Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Lotfy Makin, Doctor, Assiut University
Other Study IDs: Distance in normal ankle X-ray
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Ankle Fractures
Keywords: Radiological standard f ankle fixation
MeSH Terms: conditions — Ankle Fractures | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: X rays — Radiological assessment of vertical distance between medial and lateral malleolus in normal opulation

SUMMARY:
Determine variation in vertical distance between the medial and lateral malleolus in the normal population subjected to X-rays for any other causes than ankle fracture Determine the effect of weight bearing on this variation

DETAILED DESCRIPTION:
There is gap of knowledge about determination of vertical distance between medial and lateral malleolus Our research will cover this gap of knowledge ,so our research question will be what is the normal variation of vertical distance between medial and lateral malleolus Fractures of ankle are common injuries,approximately 2% of the general population will sustain an ankle fracture during their life time .many can be successfully treated non operatively However,for those injuries that require surgical intervention ,restoration of the anatomy is the main principle The importance of anatomic restoration of the fibula ,specially in preserving normal length has been appreciated by several authors Data will be obtained from measuring the vertical distance between lateral and medial malleolus in AP view of ankle in traumatic non ankle fractured people in standing and non standing position

ELIGIBILITY:
Inclusion Criteria:

* non ankle fractured people Non arthritic ankle Age more than 18 years old Non diabetic people Normal ankle X-rays as determined by tibiocrural angle and tibiofibular overlap

Exclusion Criteria:

* people with fracture ankle (United &non United) Arthritic ankle Diabetic people Abnormal ankle X-rays

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective cross sectional study
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Vertical distance between medial and lateral malleolus Radiologically | 1 year
  •All ankle X rays will be collected periodically through the PAC system (in Emergency Room and out patient clinics )•Using talocrural angle and tabiofibular overlapping to verify normal ankle anatomy as well as exclusion of those X rays in exclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lotfy, Study Chair — Resident of orthopedic surgery at assiut university
Locations (1):
- Michael Lotfy Makin, Asyut, Egypt